CLINICAL TRIAL: NCT01116609
Title: Local Effects of Epinephrine on Lactate, Glucose, Lipid and Protein Metabolism in Bilaterally Perfused Human Legs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: Epi-perfusion
Record Dates: First submitted 2010-04-09; First posted 2010-05-05 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: Phenylalanine; Palmitate; hyperinsulinemic-euglycemic-clamp; Effects of epinephrine in healthy volunteers
MeSH Terms: interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Epinephrine — unilateral leg infusion of Epinephrine 0.4 micrograms/m2/min
  Other Names: Adrenaline

SUMMARY:
The purpose of this study is to define the local metabolic effects of epinephrine in the bilaterally perfused human leg.

ELIGIBILITY:
Inclusion Criteria:

* Male

Exclusion Criteria:

* Comorbidity
* Females

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2004-10; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Arterio-Venous balances of metabolites | 6 hours infusion
  Acute regional effect of epinephrine infusion in the femoral artery

CONTACTS AND LOCATIONS:
Overall Officials: Niels Moller, Professor, Principal Investigator — Medical Research Laboratories, Aarhus University, Denmark
Locations (1):
- Medical research laboratories, Aarhus University Hospital, Aarhus, Denmark